CLINICAL TRIAL: NCT06979089
Title: Improving the Mental Health of Working Adults in Dutch Small and Medium-Sized Enterprises (SMEs): A Cluster RCT of WHO's Doing What Matters in Times of Stress (DWM)
Brief Title: Implementation of DWM in Dutch SMEs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Collaborators: World Health Organization (Other); University of Copenhagen (Other); University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Marit Sijbrandij, Full Professor, VU University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024.0852; ADVANCE (Other Grant/Funding Number: European Commission)
Record Dates: First submitted 2025-05-07; First posted 2025-05-18 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Anxiety; Depression; Psychological Distress
Keywords: Depression; Anxiety; Psychological Distress; Mental health; Work-place mental health; Employee well-being; Digital intervention; Online intervention; Doing What Matters in Times of Stress; Small and medium-sized enterprises
MeSH Terms: conditions — Anxiety Disorders; Depression; Psychological Well-Being; Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: The trial has cluster-randomized study design, meaning that the organizations (i.e., SMEs) that take part in the study will form clusters that will be randomized into either the intervention or control group. This way every participating employee from a SME is part of the same group.
  In this trial we are applying a stratified randomization based on whether the managers of the participating SME previously received the ASCEND intervention (manager training) or were in the control condition of a preceding trial (see NCT ID: NCT06989398). The SMEs will be randomized using limited block size that varies randomly (i.e., 4, 6, or 8 SMEs per block) per each stratum across (1) DWM and CAU (n=37) or (2) CAU only (n=37), with an equal probability of assignment to each group (allocation ratio 1:1).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doing What Matters in Times of Stress & Care-as-Usual (CAU) (Experimental): Treatment group will receive the guided-online Doing What Matters in Times of Stress (DWM) program. The program has 5 modules and is delivered in 5 weeks (one module is being made available each week).
  Treatment group also receives a weekly support call (15 minutes) from a helper (6 calls in total). Helpers are (graduate) psychology students trained according to the WHO training manual in order to provide support to participants in completing the DWM program.
  Participants in treatment group will be allowed to receive any usual care once they are enrolled in the trial.
  Interventions: Behavioral: Doing What Matters in Times of Stress
- Care-as-Usual (CAU) (No Intervention): Care-as-Usual ranges from community care to specialised psychological treatments.

INTERVENTIONS:
Behavioral: Doing What Matters in Times of Stress — DWM is the illustrated guide of the original stress management intervention - Self-Help Plus and can be offered online through a web-based application.
  DWM is a low-intensity and transdiagnostic intervention that has been designed to be widely applicable to a variety of mental health problems (depression, anxiety and PTSD). DWM is based on acceptance and commitment therapy (ACT), a modern form (third wave) of cognitive-behavioural therapy with a strong focus on mindfulness practices and identification of values, with exercises which aim to reduce distress and build social support, adaptive coping and resilience.
  DWM includes five modules, each of which focuses on a specific skill. The online version of DWM has been designed to release a module every week, so the program is finalized in 5 weeks. In this trial, participants will receive the guided version of DWM: participants will have a short (15 minutes) weekly support call with a helper (6 calls in total).
  Other Names: DWM; Doing What Matters; SH+; Self-Help Plus
  Arms: Doing What Matters in Times of Stress & Care-as-Usual (CAU)

SUMMARY:
The goal of this cluster randomized controlled trial is to explore if mental health in Dutch small and medium-sized enterprises (SMEs) can be improved by the World Health Organization's online program Doing What Matters in Times of Stress (DWM). The main questions it aims to answer are:

* Does DWM improve the mental health of employees working in Dutch SMEs?
* Does DWM improve work-related outcomes in employees working in Dutch SMEs?
* How can DWM be implemented at a large scale in Dutch SMEs?

Researchers will compare two groups to see if the DWM program is effective. One group will receive the DWM program and Care-as-Usual (group 1), and the other group will receive Care-as-Usual only (group 2).

Participants will:

* Follow the online DWM program for 5 weeks (only group 1).
* Take part in 6 telephone appointments with a facilitator (helper) that provides extra support to complete the program (only group 1).
* Complete 3 sets of questionnaires. Each set of questionnaire takes about 15 minutes to be completed (group 1 and group 2).

DETAILED DESCRIPTION:
Rationale: Small and medium-sized enterprises (SMEs) often lack the resources to combat the negative consequences of work stressors (e.g., high workplace digitalization). This puts their employees at risk of developing mental health problems. Literature on effective interventions at work for SME employees' mental health is scarce and inconclusive. This project focuses on the implementation of Doing What Matters in Times of Stress (DWM), a scalable, low-intensity, online psychological intervention developed by the World Health Organization (WHO) and adapted for use in Dutch SMEs. This study is part of the larger EU H2022-ADVANCE project, which aims to improve the mental health of vulnerable populations in Europe.

Objective: The main objective is to assess the (cost-)effectiveness of DWM in improving the mental health and work outcomes in employees of Dutch SMEs. Another objective is to identify a) barriers and facilitators to intervention engagement and adherence and b) opportunities and budget impact for scaling up the implementation of the interventions within the context of working adults in Dutch SMEs.

Study design: The first phase of this study concerns a cluster randomized controlled trial (cRCT) comparing DWM and care-as-usual (CAU) to CAU only. Main and secondary outcomes will be assessed at baseline (week 1), 1 week after completion of the 5-week intervention (week 7), and at 3-month follow-up (week 18) which is approximately 12 weeks after the end of the intervention. The second phase consists in the qualitative process evaluation that pertains individual interviews and/or focus group discussions.

Study population: In the first phase, the population is working adults in Dutch SMEs with self-reported elevated psychological distress. The aim is to include in the trial a total of 74 SMEs (37 per study arm) and to include five to 10 employees per SME (on average of seven employees; 259 per study arm, total N = 518), to detect a significant reduction in psychological distress of Cohen's d of 0.34 at 1 week post-intervention (power=0.80, two-sided alpha=0.05, ICC=0.01, 30% attrition).

In the qualitative process evaluation, the population is: participants who completed DWM and improved (n=10), who did not improve (n=10), and who dropped-out during DWM (n=10); facilitators of DWM (n=5-10); representatives of SMEs, occupational health advocacy umbrella organisations and SME umbrella organisations (n=10).

Intervention: DWM is an online intervention based on an illustrated stress management book developed by WHO. It is delivered in 5 sessions over 5 consecutive weeks, with a weekly supporting 15 minutes telephone call from a trained non-specialist facilitator (i.e., helper). DWM teaches strategies to help reduce stress such as mindfulness exercises (e.g., grounding).

Main study parameters/endpoints: The primary outcome of the cRCT will be psychological distress (combined anxiety and depression levels) at 1 week post-treatment. A decrease is anticipated in the intervention group compared to the control group, with a Cohen's d effect size of 0.34. A decrease is also anticipated in the intervention group compared to the control group in the secondary outcomes: anxiety, depression, burnout, absenteeism, presenteeism, self-stigma; and an increase in resilience, work-engagement, and quality of life Effectiveness will be assessed using linear mixed models, which account for repeated measures and clustering at the organizational/department level.

Through interviews and/or focus group discussions, the feasibility of scaling-up the implementation of the DWM intervention within the Netherlands will be examined.

ELIGIBILITY:
Inclusion Criteria (SMEs):

* Having 10 to 250 employees
* Being located in the Netherlands
* (In case of insufficient recruitment among SMEs, a mitigation strategy is to recruit individual departments from larger organizations)

Inclusion Criteria (Individual participants):

* 18 years or older
* Having elevated levels of psychological distress (Kessler Psychological Distress Scale; K10 scores > 15.9)
* Sufficient literacy and mastery (written and spoken) of one of the languages the DWM intervention is being delivered in (i.e., Dutch or English)
* Having access to an electronic device with internet access to follow the intervention
* Written informed consent before entering the study

Exclusion Criteria (Individual participants):

* Imminent suicide risk, or expressed acute needs or protection risks that require immediate follow-up
* Currently receiving specialized psychological treatment (e.g., EMDR or CBT) at the time of screening
* In case of current psychotropic medication use: being on an unstable dose for at least 2 months or a change in dosage over the past 2 months.
* Having participated in the preceding ASCEND trial as supervisor (see NCT ID: NCT06989398)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS) | Change from Baseline (week 1) to 1-week post intervention (week 7)
  The PHQ-ADS is the sum of the PHQ-9 and GAD-7 scores (details of both instruments summarised below) and thus can range from 0 to 48, with higher scores indicating higher levels of depression and anxiety symptomatology.

SECONDARY OUTCOMES:
Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS) | Change from Baseline (week 1) to 3 months follow-up (week 18)
  The PHQ-ADS is the sum of the PHQ-9 and GAD-7 scores (details of both instruments summarised below) and thus can range from 0 to 48, with higher scores indicating higher levels of depression and anxiety symptomatology.
Patient Health Questionnaire (PHQ-9) | Change from Baseline (week 1) to 1-week post intervention (week 7) and 3 months follow-up (week 18)
  PHQ-9 is a self-report measure of depression. The 9 items are scored on a 4-point scale ranging from 0 (Not at all) to 3 (Nearly every day). Scores range from 0 to 27 and higher scores indicate higher levels of depression.
Generalized Anxiety Disorder (GAD-7) questionnaire | Change from Baseline (week 1) to 1-week post intervention (week 7) and 3 months follow-up (week 18)
  GAD-7 is a self-report measure of anxiety. The 7 items are scored on a 4-point scale ranging from 0 (Not at all) to 3 (Nearly every day). Scores range from 0 to 21 and higher scores indicate higher levels of anxiety.
EQ-5D-5L | Change from Baseline (week 1) to 1-week post intervention (week 7) and 3 months follow-up (week 18)
  EQ-5D-5L is a self-report measure of quality of life. Problems experienced under 5 life domains are scored on a 5-point scale, ranging from 'No problems' to 'Extreme problems'. Higher scores indicate lower quality of life. Additionally, the current health status is measured through a visual analogue scale ranging from 'The worst health you can imagine' to 'The best health you can imagine'.
Client Service Receipt Inventory (CSRI) | Change from Baseline (week 1) to 1-week post intervention (week 7) and 3 months follow-up (week 18)
  The (mental) healthcare service utilization and related costs will be measured using the locally adapted version of the Client Service Receipt Inventory (CSRI).
Burnout Assessment Tool (BAT-4) | Change from Baseline (week 1) to 1-week post intervention (week 7) and 3 months follow-up (week 18)
  BAT-4 is a self-report measure of burnout. The 4 items are scored on a 5-point scale ranging from 1 (Never) to 5 (Always). Sores range from 1 to 5 and higher scores indicate higher levels of burnout.
Utrecht Work Engagement Scale (UWES-3) | Change from Baseline (week 1) to 1-week post intervention (week 7) and 3 months follow-up (week 18)
  UWES-3 is a self-report measure of work-engagement. The 3 items are scored on a 7-point scale ranging from 0 (Never) to 6 (Always/Every day). Scores range from 0 to 6 and higher scores indicate higher levels of work engagement.
Mainz Inventory of Microstressors (MIMIS) - adapted | Change from Baseline (week 1) to 1-week post intervention (week 7) and 3 months follow-up (week 18)
  MIMIS is a self-report measure of (micro)stressors experienced that consists of two parts.
  The first part includes three questions that measure the extent to which individuals were affected by major life events. The questions are rated on a 5-point scale, with answers ranging from from 0 (This situation did not happen) to 4 (Severe impact). Higher scores indicate a higher impact.
  The second part consists of 19 questions related to experiencing (micro)stressors which are rated on a 4-point scale, ranging from 0 (Did not happen/Almost never) to 3 ((Nearly) every day). Higher scores indicated a frequent experience of (micro)stressors.
Ultra-Brief Self-Stigma of Seeking Help Scale (SSOSH-3) | Change from Baseline (week 1) to 1-week post intervention (week 7) and 3 months follow-up (week 18)
  SSOSH-3 is a self-report measure of stigma related to mental health help-seeking behaviour. The 3 items are scored on a 5-point scale ranging from 1 (Strongly disagree) to 5 (Strongly agree). Scores range from 3 to 15. Higher scores indicate higher levels of stigma.
Absenteeism and Presenteeism | Change from Baseline (week 1) to 1-week post intervention (week 7) and 3 months follow-up (week 18)
  Absenteeism and presenteeism will be self-reported using single-item measures.
  Absenteeism: How many days have you been absent from work in the last 4 weeks due to illness?
  Presenteeism: How many days have you been less productive than usual at work in the last 4 weeks due to illness?

OTHER OUTCOMES:
Kessler-10 Psychological Distress Scale (K10) | Screening (week 1)
  K10 is a self-report measure of psychological distress. The 10 items are scored on a 5-point scale ranging from 1 (None of the time) to 5 (All of the time). Scores range from 10 to 50. Higher scores indicate higher psychological distress. In this study, the K10 is used as a screening tool, with a score greater than 15.9 indicating (at least) moderate psychological distress.
Implementation indicator: acceptability | During intervention (week 2-6)
  The implementation indicator of acceptability during the intervention (in the web-platform) will be measured for each module through one self-reported item. Answering scores range from 0 to 100, with higher scores indicating higher acceptability.
Implementation indicator: acceptability | 1-week post intervention (week 7)
  The implementation indicator of acceptability at post intervention will be measured through two self-reported items (about the program and support from helper). Answering scores range from 1 to 5, with higher scores indicating higher acceptability.
  Acceptability (alongside other relevant implementation indicators) will also be measured through qualitative interviews with participants and relevant stakeholders.
Implementation indicator: appropriateness | 1-week post intervention (week 7)
  The implementation indicator of appropriateness will be measured through one self-reported item. Answering scores range from 1 to 5, with higher scores indicating higher appropriateness.
Implementation indicator: feasibility | 1-week post intervention (week 7)
  The implementation indicator of feasibility will be measured through one self-reported item. Answering scores range from 1 to 5, with higher scores indicating higher feasibility.
Implementation indicator: barriers and facilitators | 1-week post intervention (week 7)
  The implementation indicator of barriers and facilitators will be measured through two self-reported items. Respondents are asked to identify relevant barriers and facilitators by selecting from a predefined list of response options (e.g., lack of time).
Implementation indicator: use of DWM strategies | 1-week post intervention (week 7) and 3 months follow-up (week 18)
  The implementation indicator of use of DWM strategies will be measured through three self-reported items. Respondents are asked to select the strategies they used, which they found the most useful, and to report the frequency of using the strategies, with answering scores ranging from 0 to 4. Higher scores indicate a higher usage of DWM strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Marit E. Sijbrandij, Principal Investigator — VU University of Amsterdam
Locations (1):
- Vrije Universiteit Amsterdam, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: EU-ADVANCE website — https://advancementalhealth.ku.dk/